CLINICAL TRIAL: NCT07222254
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD0292 Following Single Ascending Dose Administration to Healthy Japanese Participants
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of a Single Ascending Dose of AZD0292 in Healthy Japanese Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7700C00004
Record Dates: First submitted 2025-10-28; First posted 2025-10-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD0292 Dose Level 1 (Experimental): Participants will receive AZD0292 (dose level 1) or matching placebo on Day 1.
  Interventions: Drug: AZD0292; Drug: Placebo
- AZD0292 Dose Level 2 (Experimental): Participants will receive AZD0292 (dose level 2) or matching placebo on Day 1.
  Interventions: Drug: AZD0292; Drug: Placebo

INTERVENTIONS:
Drug: AZD0292 — Single dose of AZD0292 will be administered as an IV infusion.
Drug: Placebo — Single dose of placebo will be administered as an IV infusion.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics (PK) of single ascending doses of AZD0292 administered via intravenous (IV) infusion in healthy Japanese participants.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, placebo-controlled, single ascending dose study in healthy Japanese participants to investigate 2 dose levels of AZD0292. Participants will be randomized to receive either AZD0292 or placebo, proceeding with sentinel cohorts.

The study will comprise:

* A Screening Period of maximum 28 days.
* A Treatment Period during which participants will be resident at the site from the day before study intervention administration (Day -1) until at least 24 h post-EOI with study intervention; and discharged on Day 2.
* A Follow-up Period from Day 3 to Day 16.
* An extended Follow-up Period from Day 17 to Day 161.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese participants with suitable veins for cannulation or repeated venipuncture.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test and must not be lactating.
* Participants must agree to use an approved method of highly effective contraception as defined in the protocol.
* Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 45 kg at screening.

Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy, other than treated non-melanoma skin cancers or locally-treated cervical cancer, in the previous 5 years.
* Any clinically important illness, chronic infections or individuals who are at increased risk of infection.
* History of acquired or inherited immunodeficiency disorders.
* History of severe coronavirus disease 2019 (COVID-19) infection requiring hospitalization within the last 12 months or clinical history compatible with ongoing long COVID-19.
* Current smokers or those who have smoked or used nicotine products within the previous 6 months prior to screening.
* History of alcohol or drug abuse within the past 2 years.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD0292 and excipients contained in AZD0292.
* Known hypersensitivity to antihistamines.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs) and adverse event of special interest (AESI) | Up to Extended Follow-up Period (Day 161)
  To assess the safety and tolerability of AZD0292 following IV administration of single ascending doses to healthy Japanese adult participants.

SECONDARY OUTCOMES:
Maximum observed drug concentration (Cmax) | From Day 1 to Extended Follow-up Period (Day 161)
  To characterize the Cmax of AZD0292 following administration of single ascending doses of AZD0292 to healthy Japanese adult participants.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | From Day 1 to Extended Follow-up Period (Day 161)
  To characterize the AUClast of AZD0292 following administration of single ascending doses of AZD0292 to healthy Japanese adult participants.
Area under concentration-time curve from time 0 to infinity (AUCinf) | From Day 1 to Extended Follow-up Period (Day 161)
  To characterize the AUCinf of AZD0292 following administration of single ascending doses of AZD0292 to healthy Japanese adult participants.
Number of participants with positive anti-drug antibodies (ADAs) to AZD0292 in serum | From Day 1 to Extended Follow-up Period (Day 161)
  To evaluate the ADA responses following administration of single ascending doses of AZD0292 to healthy Japanese adult participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/